CLINICAL TRIAL: NCT03063489
Title: Evaluation of the Safety, Systemic Pharmacokinetics, and Tolerability of Single and Repeat Ocular Instillations of Loteprednol Etabonate Ophthalmic Gel, in Normal Healthy Volunteers
Brief Title: Evaluation of the Safety, Systemic Pharmacokinetics, and Tolerability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 864
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2016-12

CONDITIONS: Eye Pain
MeSH Terms: conditions — Eye Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Loteprednol Etabonate Ophthalmic Gel (Experimental): Formulated LE into a gel (loteprednol etabonate ophthalmic gel, [Lotemax® gel])
  Interventions: Drug: Loteprednol Etabonate Ophthalmic Gel

INTERVENTIONS:
Drug: Loteprednol Etabonate Ophthalmic Gel — Formulated LE into a gel (loteprednol etabonate ophthalmic gel, [Lotemax® gel])
  Other Names: LE

SUMMARY:
Evaluation of the Safety, Systemic Pharmacokinetics, and Tolerability of Single and Repeat Ocular Instillations of Loteprednol Etabonate Ophthalmic Gel, in Normal Healthy Volunteers

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the systemic pharmacokinetics (PK) of LE (loteprednol etabonate ophthalmic gel), 0.38% in normal healthy volunteer subjects at least 18 years of age and with a normal ophthalmic history. Systemic PK will be assessed in this study after a single dose and after 2 weeks of daily BID dosing.

ELIGIBILITY:
Key Inclusion Criteria:

* Are able to read, understand and provide written informed consent on an Informed Consent Form (ICF) approved by the Institutional Review Board (IRB)/Independent Ethics Committee (IEC).
* Be a non-smoking male or female at least 18 years of age on the date the ICF is signed and with the capacity to provide voluntary informed consent.
* Be in general good health and free of any concomititant conditions or treatment that could interfere with study conduct, influence the interpretation of study observations/results, or place the subject at increased risk during the study.
* Be willing/able to return for all required study visits and follow instructions from the study Investigator and his/her staff.
* Are able to self-administer eye drops or have a clinical staff member deliver the single dose of investigational product (IP) on specified study days.
* Have a normal physical examination and clinical laboratory evaluation

Key Exclusion Criteria:

* Have a history/presence of chronic generalized systemic disease that the Investigator feels might increase the risk to the subject, confound the result(s) of the study, or preclude study treatment or follow-up.
* Have any current disease or medical condition that requires medicinal therapy.
* Have a history of drug or alcohol abuse in the last 6 months.
* Have a positive urine screen for alcohol, amphetamines, barbiturates, benzodiazepines, cocaine (or cocaine metabolite), cannabinoids, methadone, methamphetamine, opiates and/or phencyclidine.
* Are known to have a prior positive blood screen for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus types 1 and 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Blood samples will be collected for the determination of loteprednol etabonate concentrations in plasma samples | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Denise Ramjit, Study Director — Valeant Pharmaceuticals
Locations (6):
- United States (6):
  - Valeant Site 01, Phoenix, Arizona
  - Valeant Site 03, Oceanside, California
  - Valeant Site 05, Miami, Florida
  - Valeant Site 04, Quincy, Massachusetts
  - Valeant Site 06, Kansas City, Missouri
  - Valeant Site 02, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes